CLINICAL TRIAL: NCT00672256
Title: Neuroimaging Decision Making and Response Inhibition During Smoking Abstinence
Acronym: SmokeAtt02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00011917; DA017261; 9270 (Other: Duke legacy protocol number)
Record Dates: First submitted 2008-05-04; First posted 2008-05-06 (Estimated); Results first posted 2013-02-15 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2013-03

CONDITIONS: Smoking
Keywords: Smoking; fMRI
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Smokers not interested in quitting smoking (Experimental): Smokers were scanned 24 hours after quitting smoking, and scanned after smoking as usual.
  Interventions: Behavioral: Smoking Abstinence

INTERVENTIONS:
Behavioral: Smoking Abstinence — Smokers were scanned after having quitting smoking for 24 hours, and scanned after smoking as usual.

SUMMARY:
The broad objective of this proposal is to identify functional neuroanatomical correlates of impairments in response inhibition during smoking abstinence. We will measure changes in performance and regional blood oxygenation levels using functional magnetic resonance imaging (fMRI)while smokers complete tasks designed to assess decision making and response inhibition.

Our primary hypothesis is that smoking abstinence will result in impaired response inhibition accompanied by decreases in blood-oxygenation-level-dependent (BOLD) fMRI signal in brain regions associated with these cognitive processes including frontal cortex and the ventral striatum. Abstinence may also result in performance-related increases in activation in brain regions associated with effortful processing including the anterior cingulate cortex in effort to compensate for deficits in other regions.

DETAILED DESCRIPTION:
Participants will learn and practice a Go/No-Go reaction time task (Garavan, Hester, Murphy, Fassbender, & Kelly, 2006) that measures inhibitory and excitatory aspects of behavioral control. During the task subjects are presented with an alternating series of Xs and Ys in the center of the screen and must press a button every time they see a Go trial (the letter 'Y' or the letter 'X') while inhibiting a response when they are presented with a No-Go trial (any interruption of the X Y alternating stream, e.g., X Y Y).

ELIGIBILITY:
Inclusion Criteria:

Smoker subjects must have

* smoked an average of 10 cigarettes per day for two continuous years of a brand that delivers (by Federal Trade Commission rated yields) at least 0.5 mg nicotine
* have an expired air carbon monoxide reading of at least 10 ppm.
* must be in general good health

Non-smoker subjects must have

* smoked less than 50 cigarettes in their lifetime
* have not smoked in the last six months
* have an expired air carbon monoxide reading of less than or equal to 5 ppm.
* must be in general good health.

Exclusion Criteria:

* major medical condition
* anything that would make participation unsafe (e.g., have pacemaker or other metallic implant) or uncomfortable (e.g., chronic pain)
* psychiatric condition
* suffering from claustrophobia
* current alcohol or drug abuse
* smokeless tobacco use, or use of nicotine replacement therapy or other smoking cessation treatment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis J McClernon, Ph.D, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: community recruitment completed recruitment March 2009
Pre-assignment Details: enrolled participants would be excluded if they were unable to meet study requirements, or had scheduling issues.
Groups:
- Smokers: Men and women ages 18-50 who smoke at least 10 cigarettes per day of a brand delivery at least 0.5 mg of nicotine for at least 2 years.
Period: Overall Study
Arm/Group | Smokers
Started | 62 (January 2007)
Completed | 18
Not Completed | 44
Not completed — PI dropped, bad data | 44

BASELINE CHARACTERISTICS:
Arm/Group | Smokers
Number analyzed (Participants) | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 62
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 35
Region of Enrollment [Number; unit: participants]
  United States | 62

OUTCOME MEASURES:

1. Primary Outcome: Signal Change in Functional Magnetic Resonance Imaging (fMRI) BOLD Signal Between Response Inhibition Trials and Control Trials in Right Inferior Frontal Cortex (rIFC) During Task on Satiated Day
Description: Percent signal change in fMRI BOLD response in rIFC to correctly inhibited targets (as compared to control trials) during a response inhibition task following smoking as usual.
  Response inhibition trials are trials in the task in which the participant must inhibit a response (not press the button)when presented with a No-Go trial. Control trials are trials in the task in which the participant must press the button when presented with a Go trial.
Time Frame: 12.5 minutes of fMRI scanning following smoking as usual
Population: 18 participants completed all aspects of the study. Two participants were excluded from analyses because they reported falling asleep in the scanner and one was excluded because of an incidental finding during the scan.
Measure: Mean (Standard Deviation); unit: percentage of signal change
Arm/Group | Smokers
Number analyzed (Participants) | 15
percentage of signal change | 0.039 (0.099)
Statistical Analysis 1: Comparison: Smokers; Within group repeated measures design. Null hypothesis is that there will be no difference in percent signal change during active task relative to baseline; Test type: Superiority or Other; p < 0.05, Paired t-test; Mean Difference (Final Values) = 0.039

2. Primary Outcome: Signal Change in fMRI BOLD Signal Between Response Inhibition Trials and Control Trials in Right Inferior Frontal Cortex (rIFC) During Task on Abstinent Day
Description: Percent signal change in fMRI BOLD response in rIFC to correctly inhibited targets (as compared to control trials) during a response inhibition task following not smoking for 24 hours.
  Response inhibition trials are trials in the task in which the participant must inhibit a response (not press the button)when presented with a No-Go trial. Control trials are trials in the task in which the participant must press the button when presented with a Go trial.
Time Frame: 12.5 minutes of fMRI scanning following 24 hrs smoking abstinence
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of signal change
Arm/Group | Smokers
Number analyzed (Participants) | 15
percentage of signal change | 0.104 (0.141)
Statistical Analysis 1: Comparison: Smokers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Paired t-test; Mean Difference (Final Values) = 0.104

3. Primary Outcome: Signal Change in fMRI BOLD Signal Between Response Inhibition Trials and Control Trials in Presupplementary Motor Area (Pre-SMA) During Task on Abstinent Day
Description: Percent signal change in fMRI BOLD response in pre-SMA to correctly inhibited targets (as compared to control trials) during a response inhibition task following not smoking for 24 hours.
  Response inhibition trials are trials in the task in which the participant must inhibit a response (not press the button)when presented with a No-Go trial. Control trials are trials in the task in which the participant must press the button when presented with a Go trial.
Time Frame: 12.5 minutes of fMRI scanning following 24 hrs smoking abstinence
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of signal change
Arm/Group | Smokers
Number analyzed (Participants) | 15
percentage of signal change | 0.173 (0.123)
Statistical Analysis 1: Comparison: Smokers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Paired t-test; Mean Difference (Final Values) = 0.173

4. Primary Outcome: Signal Change in fMRI BOLD Signal Between Response Inhibition Trials and Control Trials in Presupplementary Motor Area (Pre-SMA) During Task on Satiated Day
Description: Percent signal change in fMRI BOLD response in pre-SMA to correctly inhibited targets (as compared to control trials) during a response inhibition task following smoking as usual.
  Response inhibition trials are trials in the task in which the participant must inhibit a response (not press the button)when presented with a No-Go trial. Control trials are trials in the task in which the participant must press the button when presented with a Go trial.
Time Frame: 12.5 minutes of fMRI scanning following smoking as usual
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of signal change
Arm/Group | Smokers
Number analyzed (Participants) | 15
percentage of signal change | 0.169 (0.170)
Statistical Analysis 1: Comparison: Smokers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Paired t-test; Mean Difference (Final Values) = 0.169

ADVERSE EVENTS:
Arm/Group | Smokers
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No